CLINICAL TRIAL: NCT03788785
Title: Smoking Tobacco Cessation Integrated Program of Patients Treated for the Head and the Neck Cancer: a Controlled Randomized Study
Brief Title: Smoking Tobacco Cessation Integrated Program of Patients Treated for the Head and the Neck Cancer
Acronym: INTENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: K160704J
Record Dates: First submitted 2018-12-07; First posted 2018-12-28 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Carcinoma, Squamous Cell of Head and Neck; Tobacco Use Disorder
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: This is an open, controlled, randomized, parallel-group, two-arm, multicenter clinical study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): The specific tobacco cessation intervention of the treatment group will begin during the diagnostic phase of the HNSCC by three ½ hour session of assessment of current addictive behaviors and motivation to change smoking habits occurring within five days top. The most important point is that this intervention will be provided by trained nurses of the health care team within the ENT department, rather than in an external smoking cessation center.
  Interventions: Behavioral: Experimental arm
- Control arm (Other): In the control arm, patients will receive the current standard of care for these patients, namely referral to external care after general advice on tobacco cessation (self-help tools).
  Interventions: Other: Control arm

INTERVENTIONS:
Behavioral: Experimental arm — The specific tobacco cessation intervention will be based on meeting with trained nurses : three 1/2 hour session of assessment of current addictive behaviors and motivation to change smoking habits occurring within five days tops.
  Other Names: Specific tobacco cessation intervention
  Arms: Experimental arm
Other: Control arm — In the control arm, patients will receive the current standard of care for these patients, namely referral to external care after general advice on tobacco cessation (self-help tools).
  Other Names: Standard tobacco cessation intervention
  Arms: Control arm

SUMMARY:
Head and neck squamous cell carcinomas (HNSCCs) arise in the mucosa of the upper aero-digestive tract. They are the 6th most prevalent type of cancer worldwide. The risk related to tobacco is particularly high in the case of HNSCC, as the prevalence of heavy smoking for long periods is high in this population. The investigators' aim is to compare two models: one is a specific model of tobacco cessation intervention designed for health care teams treating patients with HNSCC; the other is the current standard of care for these patients, namely referral to external care after general advice on tobacco cessation. The investigators will evaluate the efficacy of this intervention 12 months after randomization. This intervention will be implemented into otolaryngology (ENT) care by training ENT nurses with a specific program for tobacco cessation delivered to patients diagnosed with HNSCC.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinomas (HNSCCs) arise in the mucosa of the upper aero-digestive tract. They are the 6th most prevalent type of cancer worldwide, with approximately 600 000 new cases every year. The investigators hypothesize that a specifically-designed tobacco cessation intervention initiated and driven by trained nurses of the health care team, either in the otolaryngology (ENT) department or in the radiotherapy department, is more efficient than a classic intervention based on the same pharmacological support during the hospital stay (NRT) followed by an orientation in an external smoking cessation center, while remaining feasible for both patients and caregivers.The health care setting represents an ideal place to initiate cessation interventions with smokers who are newly diagnosed with a malignancy. The investigators' aim is to compare two models: one is a specific model of tobacco cessation intervention designed for health care teams treating patients with HNSCC; the other is the current standard of care for these patients, namely referral to external care after general advice on tobacco cessation. The investigators will evaluate the efficacy of this intervention 12 months after randomization. This intervention will be implemented into otolaryngology (ENT) care by training ENT nurses with a specific program for tobacco cessation delivered to patients diagnosed with HNSCC.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Patients diagnosed with HNSCC and oriented toward any combination of the following treatment: surgery, radiotherapy within one of the study sites, chemotherapy
3. Patient who smoked in the last 3 months
4. Negative pregnancy test for women of childbearing age
5. For men and women : Using effective contraceptive methods during treatment and within 3 months after the end of treatment for men with her partner of childbearing age
6. Having signed written informed consent

Exclusion Criteria:

1. Patient's refusal to participate
2. Life expectancy <6 months defined by multidisciplinary staff
3. Lack health insurance (French social security)
4. Current guardianship
5. Non French-speaking patient
6. Living outside catchment area (200 kM around North Paris)
7. Severe cognitive impairment or unstable medical condition (psychiatric or other) that does not permit informed consent and/or continuation of the questionnaire
8. Pregnancy, breastfeeding or lack of appropriate contraception during study duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Smoking abstinence | at 12 months after randomization
  Proportion of patients with continuous abstinence during the last 6 months of the study, defined as having negative cotinine urine test at the last three visits.

SECONDARY OUTCOMES:
Reduction of Tobacco consumption | 12 months
  Proportion of patients with a 50% reduction or more of tobacco consumption between endpoint and baseline
Reduction of Nicotine dependance | 12 months
  Proportion of patients with a 50% reduction or more at the Heaviness of Smoking Index (HSI) score between endpoint and Baseline. The Heavy smoking index (HSI) is the combination of two items (each scored between 0 and 3). The score range from 0 to 6. The cut-off point is 4. A high HSI score defined by a score of 4 or higher indicated high nicotinine dependance.
Proportion of patients with at least one visit with negative cotinine urine test | 12 months
Tolerance of cancer treatments | at 2 months
  Proportion of reduction of adverse events reported
Tolerance of cancer treatments | at 4 months
  Proportion of reduction of adverse events reported
Tolerance of cancer treatments | at 6 months
  Proportion of reduction of adverse events reported
Tolerance of cancer treatments | at 8 months
  Proportion of reduction of adverse events reported
Tolerance of cancer treatments | at 10 months
  Proportion of reduction of advrese events reported
Tolerance of cancer treatments | at 12 months
  Proportion of reduction of adverse events reported
Satisfaction evaluated on a custom questionnaire | at 12 months
  Good satisfaction, feasibility and transferability of the intervention felt reported nurses on a custom questionnaire.
Psychological state | at 12 months
  Decrease in Hospital Anxiety and Depression scale (HAD) mean scores over time.
  The HAD scale is a self-assessment scale for detecting states of depression and anxiety in the setting of an hospital medical outpatient clinic.
  HADS is a self-administered scale of 14 items which assessed levels of depression and anxiety, divided into 2 subscales of 7 items (Anxiety or HADS-A, Depression or HADS-D). Each item is scored on a scale of 0 to 3. A score is generated for each of the two sub-scales (sum of the 7 items, ranging from 0 to 21). Limit scores, for each of the scores, distinguish: non-cases or asymptomatic ones (score ≤ 7); probable or borderline cases (score 8-10); clearly or clinically symptomatic cases (score ≥ 11).
Quality of life evaluated using the Euro-Quality of life - 5 Dimensions (EQ5D) scale | at 2 months
  The EQ-5D-5L is composed of - the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Each level corresponds to 1-digit number expressing the level selected for that dimension.
  The EQ VAS corresponds to a 20 cm vertical, visual analogue scale raging from 'the best health you can imagine' to 'the worst health you can imagine'.
Quality of life evaluated using the Euro-Quality of life - 5 Dimensions (EQ5D) scale | at 4 months
  The EQ-5D-5L is composed of - the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Each level corresponds to 1-digit number expressing the level selected for that dimension.
  The EQ VAS corresponds to a 20 cm vertical, visual analogue scale raging from 'the best health you can imagine' to 'the worst health you can imagine'.
Quality of life evaluated using the Euro-Quality of life - 5 Dimensions (EQ5D) scale | at 6 months
  The EQ-5D-5L is composed of - the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Each level corresponds to 1-digit number expressing the level selected for that dimension.
  The EQ VAS corresponds to a 20 cm vertical, visual analogue scale raging from 'the best health you can imagine' to 'the worst health you can imagine'.
Quality of life evaluated using the Euro-Quality of life - 5 Dimensions (EQ5D) scale | at 8 months
  The EQ-5D-5L is composed of - the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Each level corresponds to 1-digit number expressing the level selected for that dimension.
  The EQ VAS corresponds to a 20 cm vertical, visual analogue scale raging from 'the best health you can imagine' to 'the worst health you can imagine'.
Quality of life evaluated using the Euro-Quality of life - 5 Dimensions (EQ5D) scale | at 10 months
  The EQ-5D-5L is composed of - the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Each level corresponds to 1-digit number expressing the level selected for that dimension.
  The EQ VAS corresponds to a 20 cm vertical, visual analogue scale raging from 'the best health you can imagine' to 'the worst health you can imagine'.
Quality of life evaluated using the Euro-Quality of life - 5 Dimensions (EQ5D) scale | at 12 months
  The EQ-5D-5L is composed of - the EQ-5D-5L descriptive system and the EQ Visual Analogue scale (EQ VAS). The descriptive system comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Each level corresponds to 1-digit number expressing the level selected for that dimension.
  The EQ VAS corresponds to a 20 cm vertical, visual analogue scale raging from 'the best health you can imagine' to 'the worst health you can imagine'.
Pain assessed by pain-killer consumption | at 2 months
  Decreased cumulated pain-killer consumption at each visit (morphine-equivalent)
Pain assessed by pain-killer consumption | at 4 months
  Decreased cumulated pain-killer consumption at each visit (morphine-equivalent)
Pain assessed by pain-killer consumption | at 6 months
  Decreased cumulated pain-killer consumption at each visit (morphine-equivalent)
Pain assessed by pain-killer consumption | at 8 months
  Decreased cumulated pain-killer consumption at each visit (morphine-equivalent)
Pain assessed by pain-killer consumption | at 10 months
  Decreased cumulated pain-killer consumption at each visit (morphine-equivalent)
Pain assessed by pain-killer consumption | at 12 months
  Decreased cumulated pain-killer consumption at each visit (morphine-equivalent)
Treatment response | at 2 months
Treatment response | at 4 months
Treatment response | at 6 months
Treatment response | at 8 months
Treatment response | at 10 months
Treatment response | at 12 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Lariboisiere hospital, Paris
  - Bichat hospital, Paris
  - Tenon hospital, Paris

IPD SHARING:
Plan to Share IPD: Undecided